CLINICAL TRIAL: NCT05746416
Title: Xience Registry Study for the Impact of Early Use of Low-Dose Ticagrelor-Based Dual Antiplatelet Therapy to Clinical Outcomes in Patient Undergoing Percutaneous Coronary Interventions for Complex Lesions
Brief Title: Xience Registry In Complex Lesion of Acute Coronary Syndrome Patients witH Ticagrelor (RICH)
Acronym: RICH
Status: Completed | Type: Observational
Sponsor: Hanyang University Seoul Hospital (Other)
Collaborators: Soon Chun Hyang University (Other); Abbott (Industry)
Responsible Party: Principal Investigator, Young-Hyo Lim, professor, Hanyang University Seoul Hospital
Other Study IDs: RICH_2020-0104
Record Dates: First submitted 2023-02-13; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention; Acute Coronary Syndrome
Keywords: Low-dose ticagrelor-based dual antiplatelet agent therapy; Percutaneous coronary intervention; Acute coronary syndrome; Complex coronary lesion; Net clinical outcome; Everolimus-eluting stent
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- s-TDAPT group: Ticagrelor 180mg + Aspirin 100mg within 6 months after index PCI
- l-TDAPT group: Ticagrelor 120mg + Aspirin 100mg within 6 months after index PCI

SUMMARY:
The goal of this multicenter prospective clinical cohort study is to investigate the impact of early use of low-dose Ticagrelor-based dual antiplatelet agent therapy (TDAPT) (ticagrelor 120mg daily; l-TDAPT) as compared to standard-dose TDAPT (ticagrelor 180mg daily; s-TDAPT) in outcomes of percutaneous coronary intervention (PCI).

The main question it aims to answer are:

Given the low ischemic risk and high bleeding tendency in Asians, the low dose TDAPT may provide better net clinical benefits of ischemic and bleeding events than the standard dose TDAPT.

DETAILED DESCRIPTION:
Participants were administrated with 300mg of Aspirin and 180mg of ticagrelor orally before they underwent index PCI, and were prescribed with s-TDAPT from the next day after index PCI at least for 1 week. The start of l-TDAPT was decided by each attending physician's preference.

Successful PCI was defined as a residual stenosis <30% with Thrombolysis in Myocardial Infarction grade 3 flow after PCI and the absence of death by MI and reintervention for the index coronary lesions during the admission period. Standard definitions of cardiovascular events were used for all clinical events. Myocardial infarction (MI) was defined using the 4th universal definition of MI as previously described. Repeat revascularization (RR) was defined as a new PCI for the target vessels or de-novo coronary lesions. All-cause death was defined as a death from any cause. Cardiovascular death was defined as death from MI, stent thrombosis and ischemic stroke. A major adverse cardiac and cerebrovascular event (MACE) was defined as a composite of cardiovascular death, non-fetal MI, RR, stent thrombosis and ischemic stroke. A bleeding event was defined as the bleeding event equivalent to Bleeding Academic Research Consortium (BARC) classification 2 or higher. A net clinical event (NCE) was defined as a composite of MACEs and bleeding events. Patients were scheduled to follow up to 2 years after index PCI. Clinical follow-up started when a patient discharged from the hospitalization for the index PCI and ended when the patient experienced the any clinical event or reached the end of follow-up. The follow-up visits were scheduled at 1, 3 and 6 months, 1 year and 2 years after discharge.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* acute coronary syndrome (ACS) undergoing PCI
* PCI for complex coronary lesions using everolimus-eluting stents (Xience®, Abbot corp, Chicago, Illinois, US)
* prescribed with s-TDAPT for more than 3 months

Exclusion Criteria:

* cardiogenic shock
* PCI using drug-eluting stents (DES) other than the everolimus-eluting stents
* those who had conditions requiring a long-term oral anticoagulant therapy
* those with life expectancy <1 year

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 19 years of age or older with acute coronary syndrome (ACS) undergoing PCI for complex coronary lesions using everolimus-eluting stents (Xience®, Abbot corp, Chicago, Illinois, US) and prescribed with s-TDAPT were enrolled in the registry. The enrollment was decided after a patient had undergone PCI and before the patient was discharged from the PCI center
Sampling Method: Non-Probability Sample
Enrollment: 977 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
A major adverse cardiac and cerebrovascular event (MACE) | at 1 years after discharge
  a composite of cardiovascular death, non-fetal MI, RR, stent thrombosis and ischemic stroke.

SECONDARY OUTCOMES:
All cause death | at 1 years after discharge
  a death from any cause
cardiovascular death | at 1 years after discharge
  death from MI, stent thrombosis and ischemic stroke
Myocardial infarction | at 1 years after discharge
  the 4th universal definition of MI
Repeat revascularization | at 1 years after discharge
  a new PCI for the target vessels or de-novo coronary lesions
bleeding event | at 1 years after discharge
  the bleeding event equivalent to Bleeding Academic Research Consortium (BARC) classification 2 or higher
A net clinical event (NCE) | at 1 years after discharge
  a composite of MACEs and bleeding events

CONTACTS AND LOCATIONS:
Locations (1):
- Young-Hyo Lim, Seoul, South Korea